CLINICAL TRIAL: NCT03666637
Title: The Relationship Between Femoral Neck Fracture in Adult and Avascular Necrosis and Nonunion
Brief Title: Femoral Neck Fracture in Adult and Avascular Necrosis and Nonunion
Status: Completed | Type: Observational
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, Raheef Alatassi, Orthopedic Surgeon, Security Forces Hospital
Other Study IDs: femoral neck fracture in adult
Record Dates: First submitted 2018-09-08; First posted 2018-09-12 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Femoral Neck Fractures; Avascular Necrosis
Keywords: Adult; avascular necrosis; Complications; Delayed fixation; nonunion; Surgical timing; Pauwels
MeSH Terms: conditions — Femoral Neck Fractures; Osteonecrosis | interventions — deoxyhypusine synthase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: dynamic hip screw (DHS) and cannulated screw (CS) — A preformed case report form was used to collect the data which included the demographic profile of the patients (age, gender), comorbidities, smoking history, mode of injury (high or low energy), presence of multiple trauma, garden classification, side of injury, time to fixation (in hours), type of reduction, type of implant used, RUSH score (healing), start of weight bearing, development of AVN, and final outcome (whether varus, valgus, displaced or healed).
  Other Names: Time to fixation

SUMMARY:
One of the most serious sequelae of femoral neck fractures (FNFs) is avascular necrosis (AVN) and nonunion, and this translates to a significant morbidity and mortality. This study was conducted to determine the relationship between the etiologies and management of FNFs in our institution and its relationship to the development of AVN or nonunion.

DETAILED DESCRIPTION:
Femoral neck fractures (FNFs) are fractures of the flattened pyramidal bone connecting the femoral head and the femoral shaft. It is not so common in healthy individuals but common among athletes, military recruits, and young adults because of high energy cases such as sports and road traffic accidents, in adults due to falls, in women with estrogen imbalances, and in patients with bone mineralization and deficiencies.

In the USA in 2013, there were a reported 146 cases per 100,000 population. Mortality can be high as much as 30% at one year particularly if there is delaying management over 24 hours.

FNFs are classified using the Garden Classification based on anteroposterior radiographs into Types I to IV wherein Type I is incomplete fracture, Type II is complete but non-displaced fracture, Type III is complete and partially displaced fracture and Type IV is complete and fully displaced femur. Another classification is the Pauwel's classification which is a biomechanical classification based on the vertical orientation of the fracture line, and is commonly used to determine the appropriate treatment for FNFs particularly among younger adults.

The radiographic union score for hip (RUSH) is a scoring used to describe healing of femoral neck fractures, particularly among patients who might require additional surgery, in which patients with a 6-month RUSH score <18 have a greater probability of undergoing reoperation.

Surgical management of FNFs include open reduction and internal fixation (ORIF) which has some fixation failures, primary total hip arthroplasty (TA) which is cost-effective for displaced FNFs in patients 45-65 years old, cannulated screw (CS) fixation for the young and middle-aged patients, dynamic hip screw fixation (DHS), and hemiarthroplasty. The decision to use either of the surgical management depends on several factors including displacement of the femoral neck, presence of hip joint arthritis, age, and other factors. Around 24% of patients who had THA underwent revision within 5 years because of aseptic loosening, infection and many other causes. Some surgeons however prefer ORIF and some prefer THA for displaced FNFs particularly among active older patients with Garden III fracture.

One of the most serious sequelae of FNFs is avascular necrosis (AVN) which occurs in 10-45% of patients with FNFs, particularly those who have displaced and nonunion FNFs. Nonunion occurs in almost 20% of FNFs, more common in men than women, and common with increasing age. Around 33% of displaced FNFs are associated with complications. One study showed that age and the type of fixation are not significantly correlated to the incidence of AVN, but the amount of vascular damage at the time of the fracture determines the development of vascular necrosis. On the other hand, a separate study showed that the fracture type and age are the most significant predictors of the development of AVN.

It has been mentioned that time is essential in the management of FNFs particularly in the development of AVN. One study showed that the rates of AVN increases over time when patients underwent surgery before 12 hours had elapsed and after 12 hours from 12.5% to 14.0%, while another study showed that a delay of more than 48 hours before surgery did not influence the rate of union or the development of AVN when compared with operation within 48 hours of injury. Some studies reported that bleeding from the holes of cannulated screws predict the development of AVN, some due to damage to the blood supply of the femoral head brought about by the initial high energy trauma, and some due to the extent of fracture displacement. Other studies have suggested that FNFs treated using cannulated screws particularly among middle-aged and elderly patients have less incidence of AVN. Because of these, we undertook this study to determine the relationship between the etiologies and management of FNFs in our institution and its relationship to the development of AVN or nonunion.

ELIGIBILITY:
Inclusion Criteria:

* All patients included must be adult and aged 18 years old to 70 years old
* admitted and managed for Femur Neck Fracture.
* All fresh trauma and referred cases were included in the study.

Exclusion Criteria:

* Patients who have sickle cell disease (SCD), patients who are on steroids, patients who have developmental dysplasia of the hip (DDH), patients who have ipsilateral femoral shaft fracture, immobilized patients, pediatric cases and comatose patients were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * All adult patients aged 18 years old to 70 years old admitted and managed for Femur Neck Fracture during the last 10 years (2007 - 2017) at Security Forces Hospital, Riyadh, Saudi Arabia.
  * Fresh trauma case including all patients admitted within 24 hours of the injury.
  * Referred cases including patients referred from other hospitals and patients came from the war zone without time limitation.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of AVN in adult patients with FNF that treated surgically | Baseline
  In relation to the time of surgery after the fracture
RUSH score (healing) | 6 months
  The radiographic union score for hip (RUSH) is a scoring used to describe healing of femoral neck fractures, particularly among patients who might require additional surgery, in which patients with a 6-month RUSH score <18 have a greater probability of undergoing reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Koaban, FRCS, Study Director — Security Forces Hospital
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Kemmler W, von Stengel S, Kohl M. Exercise Frequency and Fracture Risk in Older Adults-How Often Is Enough? Curr Osteoporos Rep. 2017 Dec;15(6):564-570. doi: 10.1007/s11914-017-0407-7. PMID 28975497
- [Background] Neubauer T, Brand J, Lidder S, Krawany M. Stress fractures of the femoral neck in runners: a review. Res Sports Med. 2016 Jul-Sep;24(3):185-99. doi: 10.1080/15438627.2016.1191489. Epub 2016 Jun 6. PMID 27265356
- [Background] Morrissey N, Iliopoulos E, Osmani AW, Newman K. Neck of femur fractures in the elderly: Does every hour to surgery count? Injury. 2017 Jun;48(6):1155-1158. doi: 10.1016/j.injury.2017.03.007. Epub 2017 Mar 6. PMID 28325670
- [Background] Kazley JM, Banerjee S, Abousayed MM, Rosenbaum AJ. Classifications in Brief: Garden Classification of Femoral Neck Fractures. Clin Orthop Relat Res. 2018 Feb;476(2):441-445. doi: 10.1007/s11999.0000000000000066. No abstract available. PMID 29389800
- [Background] Shen M, Wang C, Chen H, Rui YF, Zhao S. An update on the Pauwels classification. J Orthop Surg Res. 2016 Dec 12;11(1):161. doi: 10.1186/s13018-016-0498-3. PMID 27955672
- [Background] Frank T, Osterhoff G, Sprague S, Garibaldi A, Bhandari M, Slobogean GP; FAITH Investigators. The Radiographic Union Score for Hip (RUSH) Identifies Radiographic Nonunion of Femoral Neck Fractures. Clin Orthop Relat Res. 2016 Jun;474(6):1396-404. doi: 10.1007/s11999-015-4680-4. PMID 26728521
- [Background] Hu X, Liu BJ, Wen XM, Zheng YH, Jia K. [Clinical observation of closed reduction and compression cannulated screw fixation for the treatment of femoral neck fracture in young and middle-aged patients]. Zhongguo Gu Shang. 2018 Feb 25;31(2):111-114. doi: 10.3969/j.issn.1003-0034.2018.02.003. Chinese. PMID 29536678
- [Background] Chen C, Yu L, Tang X, Liu MZ, Sun LZ, Liu C, Zhang Z, Li CZ. Dynamic hip system blade versus cannulated compression screw for the treatment of femoral neck fractures: A retrospective study. Acta Orthop Traumatol Turc. 2017 Oct;51(5):381-387. doi: 10.1016/j.aott.2017.07.006. Epub 2017 Aug 26. PMID 28844681
- [Background] Calandruccio RA, Anderson WE 3rd. Post-fracture avascular necrosis of the femoral head: correlation of experimental and clinical studies. Clin Orthop Relat Res. 1980 Oct;(152):49-84. PMID 7438624
- [Background] Karaeminogullari O, Demirors H, Atabek M, Tuncay C, Tandogan R, Ozalay M. Avascular necrosis and nonunion after osteosynthesis of femoral neck fractures: effect of fracture displacement and time to surgery. Adv Ther. 2004 Sep-Oct;21(5):335-42. doi: 10.1007/BF02850038. PMID 15727403
- [Background] Upadhyay A, Jain P, Mishra P, Maini L, Gautum VK, Dhaon BK. Delayed internal fixation of fractures of the neck of the femur in young adults. A prospective, randomised study comparing closed and open reduction. J Bone Joint Surg Br. 2004 Sep;86(7):1035-40. doi: 10.1302/0301-620x.86b7.15047. PMID 15446534